CLINICAL TRIAL: NCT01293409
Title: Transcranial Brain-Targeted Bright Light Treatment Via Ear Canals in Seasonal Affective Disorder (SAD) - a Randomized Placebo Controlled Dose Finding Study
Brief Title: Bright Light Therapy in Seasonal Affective Disorder (SAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); ODL Terveys Oy (Unknown); Valkee Oy (Industry); University of Eastern Finland (Other)
Responsible Party: Professor Pirkko Räsänen, M.D., Ph.D., University of Oulu, Institute of Clinical Medicine, Department of Psychiatry, Box 5000, FIN-90014 University of Oulu, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FI (FWA00000190) 11/2008b
Record Dates: First submitted 2011-01-21; First posted 2011-02-10 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Seasonal Affective Disorder
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): The amount of photic energy of light is considered to be non-therapeutical
  Interventions: Other: Transcranial Brain-Targeted Bright Light Treatment
- Intermediate dose (Experimental): The amount of photic energy of bright light is considered to be "intermediate"
  Interventions: Other: Transcranial Brain-Targeted Bright Light Treatment
- High dose bright light (Experimental): The amount of photic energy of bright light is considered to be fully therapeutic
  Interventions: Other: Transcranial Brain-Targeted Bright Light Treatment

INTERVENTIONS:
Other: Transcranial Brain-Targeted Bright Light Treatment — Transcranial Brain-Targeted Bright Light Treatment via Ear Canals
  Other Names: VALKEE

SUMMARY:
Bright light therapy (BLT) is widely accepted as first-line treatment of seasonal affective disorder (SAD). However, the mechanism of action of BLT is still widely unknown. On the other hand, in mammals, light penetrates the skull bone and reaches the brain, and extra ocular transcranial phototransduction has physiological influences such as changed reproductive cycles and increased brain serotonin levels. Therefore, the investigators run a randomized, placebo controlled, double blind, dose finding study on the putative effect of transcranial bright light in the treatment of SAD.

ELIGIBILITY:
Inclusion Criteria:

• a patient has (according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision [DSM-IV-TR]) a Major depression, recurrent episode, seasonal pattern, "moderate" or "severe" (classification code 296.32 and 296.33)

The 29-item Structured Interview Guide for Hamilton Depression Rating Scale - Seasonal Affective Disorder Version (SIGH-SAD) score ≥ 20

* The 29-item Structured Interview Guide for Hamilton Depression Rating Scale - Seasonal Affective Disorder Version (SIGH-SAD) score ≥ 20
* The 21-item Hamilton Depression Rating Scale score ≥ 10
* The 8-item atypical symptom score ≥ 5

  * patient is over 18 years
  * patient can read and understand the subject information sheet
  * patient has signed the informed consent form
  * patient is not pregnant

Exclusion Criteria:

* patient has a lifetime psychotic disorder
* patient has a DSM-IV Axis I disorder other than some anxiety disorder evaluated by MINI
* patient has some DSM-IV-TR Axis II disorder, which is likely to interfere with the study treatment according to the investigator
* patient has alcohol or some other substance use dependence or misuse
* patients has some unstable somatic disorder
* patient uses some psychotropic agencies
* patient is, in the opinion of the investigator, unsuitable for any reason
* patient is a member of the site personnel or their immediate families
* patient has had bright light therapy via ear canals during the current episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The 29-item Structured Interview Guide for Hamilton Depression Rating Scale - Seasonal Affective Disorder Version (SIGH-SAD) total score ≤ 8 | At the end of the four-week study period
  Remission, i.e., the 29-item Structured Interview Guide for Hamilton Depression Rating Scale - Seasonal Affective Disorder Version (SIGH-SAD) total score ≤ 8

SECONDARY OUTCOMES:
≥ 50 % decrease of the severity of symptoms as assessed by SIGH-SAD | At the end of the four-week study period
≥ 50 % decrease of the severity of symptoms as assessed by the 14-item Hamilton Anxiety Rating Scale total score | At the end of the four-week study period
≥ 50 % decrease of the severity of symptoms as assessed by the 21-item Beck depression Inventory (BDI-21) total score | At the end of the four-week study period
≥ 50 % decrease of the severity of symptoms as assessed by 21-item Hamilton Depression Rating Scale total score | At the end of the four-week study period
A number of participants with bright light therapy related (according to physician decision) adverse events as a measure of safety and tolerability | During the four week study period

CONTACTS AND LOCATIONS:
Overall Officials: Pirkko Räsänen, M.D., Ph.D., Principal Investigator — Professor
Locations (1):
- ODL Terveys Oy, Oulu, Finland

REFERENCES:
- [Derived] Jurvelin H, Takala T, Nissila J, Timonen M, Ruger M, Jokelainen J, Rasanen P. Transcranial bright light treatment via the ear canals in seasonal affective disorder: a randomized, double-blind dose-response study. BMC Psychiatry. 2014 Oct 21;14:288. doi: 10.1186/s12888-014-0288-6. PMID 25330838